CLINICAL TRIAL: NCT01799980
Title: Evaluation of Endobronchial Ultrasound (EBUS) for Staging Lung Cancer
Acronym: EBUS
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2009471-01H
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Lung Cancer
Keywords: Lung cancer; Cervical mediastinoscopy; Endobronchial ultrasound; Staging
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cervical mediastinoscopy: This group will undergo cervical mediastinoscopy before surgery to stage their lung cancer (procedure decided by the surgeon).
- Endo-bronchial ultrasound: This group will undergo endobronchial ultrasound before surgery to stage their lung cancer (procedure decided by the surgeon).

SUMMARY:
This study will compare two different methods of staging lung cancer to determine whether endobronchial ultrasound (EBUS) staging of mediastinal lymph nodes will provide good diagnostic yield in detecting lung cancer, when compared to current methods of a staging bronchoscopy and cervical mediastinoscopy.

ELIGIBILITY:
Inclusion Criteria:

Patients, > 18 years of age,

Gender- Males and Female

Diagnosis of Non Small Cell Lung Cancer.

Patients who have consented on an Ottawa Hospital consent form to undergo a mediastinoscopy procedure or EBUS-TBNA, and a Positron emission tomography (PET) of the chest for lung cancer staging.

Exclusion Criteria:

Females who are pregnant (or found to be pregnant) during the course of this research study.

Patients who do not provide their Ottawa Hospital consent to undergo a staging bronchoscopy , cervical mediastinoscopy or EBUS-TBNA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a staging procedure for lung cancer (either cervical mediastinoscopy or endobronchial ultrasound).
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2012-06; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Lung cancer staging | Pre-op and post-op
  Lung cancer staging (assessed by either cervical mediastinoscopy or EBUS) will be compared both pre-op and post-op.

CONTACTS AND LOCATIONS:
Overall Officials: Donna E Maziak, MD, MSc, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada